CLINICAL TRIAL: NCT01661023
Title: A Multidisciplinary Study of Breast Cancer in Ghana
Brief Title: The Ghana Breast Health Study
Status: Completed | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999912174; 12-C-N174
Record Dates: First submitted 2012-08-07; First posted 2012-08-09 (Estimated); Last update posted 2020-04-20 (Actual); Status verified 2020-04

CONDITIONS: Breast Neoplasms
Keywords: Breast Cancer; Epidemiology
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Background:

- Breast cancer is becoming more common in Africa. A higher number of cases appear in women under age 35 than in the developed world. However, little is known about the factors that may contribute to breast cancer in Africa. Researchers want to collect information from female patients in teaching hospitals in Accra and Kumasi, Ghana and to compare this information with that obtained from healthy women in the general population. These two hospitals treat most breast cancers in Ghana. The data will provide information regarding factors that predispose to the development of breast cancer among women in Ghana.

Objectives:

- To identify and study breast cancer risk factors in women in Ghana.

Eligibility:

* Women between 18 and 74 years of age who are diagnosed with breast cancer.
* Participants will come from teaching hospitals in Accra and Kumasi, Ghana. Women without breast cancer will be identified from the 2010 Ghanaian Census for comparison purposes

Design:

* Participants will answer questions about their health and lifestyle.
* Height, weight, and waist/hip measurements will be collected.
* Blood and saliva samples will be collected.
* Participants will be given a collection kit to collect a stool sample.
* Treatment will not be provided as part of this study.

DETAILED DESCRIPTION:
Breast cancer is becoming a more common disease in Africa, with a high proportion of cases developing among women under age 50. Despite this, there is scant information on predisposing factors in African populations. We are proposing a multidisciplinary case-control study at three hospitals in Accra and Kumasi that treat the majority of breast cancers in Ghana. We have begun this investigation as a pilot endeavor and are seeking approval for continuation into a full-scale effort, which over the two years following the pilot will result in a total of approximately 2,000 interviewed cases and 2,000 population controls. Tumor tissue samples are being sought from cases in order to classify them into subtypes (including triple negative tumors, which predominate among young African women). A detailed questionnaire is being administered in hospital and anthropometry measurements are being taken. Additionally, subjects are being asked to donate blood, saliva, and stool samples for assessment of genetic and other biologic markers. Similar materials are being collected from population controls. In addition to providing unique data relevant for improving prevention activities, this study will build capacity for additional research activities in Ghana.

ELIGIBILITY:
* ELIGIBILITY CRITERIA:

Eligible for inclusion as cases in this study will be women 18-74 years of age who have been residents of defined catchment areas surrounding the two cities for at least one year s time and who are either diagnosed at the study hospitals within the past year (KBTH, KATH, and PLH) or referred there for clinical care. The catchment area in Accra will consist of 10 districts in Greater Accra (Accra Metropolitan, Adenta, Tema, Ashaiman, Ga East, Ga West, Ledzokuku-Krowor, Weija (Ga South), Dangbe East, Dangbe West), two in the Eastern region (Suhum Kraboa Coaltar, Akwapim South) and one in the Central region (Awutu Senya). In Kumasi, the catchment area will consist of 7 districts surrounding KATH and PLH (Atwima Kwanwoma, Atwima Nwabiagya, Bosumtwi, Ejisu Juaben, Afigya Kwabre, Kwabre, and Kumasi Metropolitan).

Ages: 18 Years to 74 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The source of breast cancer cases included the two largest teaching/cancer treatment hospitals in the country, Korle Bu Teaching Hospital in Accra and Komfo Anoyke Teaching Hospital in Kumasi, as well as Peace and Love Hospital, a private hospital in Kumasi that specializes in breast cancer care and diagnoses and treats a large number of breast cancer patients. Eligibility criteria for study cases included being recommended for a biopsy given lesions suspicious of malignancy or presenting at a @@@study hospital for treatment of pathologically documented breast cancers diagnosed within the preceding year.Controls were selected from women in the catchment area of the hospitals using data from the 2010 Census, matched on age and geographical area to the the cases.@@@@@@
Sampling Method: Probability Sample
Enrollment: 4241 (Actual)
Dates: Start 2012-07-19 (Actual); Primary Completion 2016-04-25 (Actual); Study Completion 2020-04-16 (Actual)

PRIMARY OUTCOMES:
Breast Cancer | Within one year of diagnosis
  Pathologically confirmed diagnosis of breast cancer

SECONDARY OUTCOMES:
Benign breast disease | At biopsy

CONTACTS AND LOCATIONS:
Overall Officials: Montserrat Garcia-Closas, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (2):
- Ghana (2):
  - University of Ghana, Accra
  - Kwane Nkrumah University of Science and Technology, Kumasi

REFERENCES:
- [Background] Huo D, Ikpatt F, Khramtsov A, Dangou JM, Nanda R, Dignam J, Zhang B, Grushko T, Zhang C, Oluwasola O, Malaka D, Malami S, Odetunde A, Adeoye AO, Iyare F, Falusi A, Perou CM, Olopade OI. Population differences in breast cancer: survey in indigenous African women reveals over-representation of triple-negative breast cancer. J Clin Oncol. 2009 Sep 20;27(27):4515-21. doi: 10.1200/JCO.2008.19.6873. Epub 2009 Aug 24. PMID 19704069
- [Background] Akarolo-Anthony SN, Ogundiran TO, Adebamowo CA. Emerging breast cancer epidemic: evidence from Africa. Breast Cancer Res. 2010 Dec 20;12 Suppl 4(Suppl 4):S8. doi: 10.1186/bcr2737. No abstract available. PMID 21172092
- [Background] Walker AR, Adam FI, Walker BF. Breast cancer in black African women: a changing situation. J R Soc Promot Health. 2004 Mar;124(2):81-5. doi: 10.1177/146642400412400212. PMID 15067980